CLINICAL TRIAL: NCT02191384
Title: Proof Of Concept Study of Orcinoside in the Treatment of Major Depressive Disorder(MDD): a Randomized, Double-Blind, Placebo-Paralleled,Dose-Finding, Multicenter Clinical Trial
Brief Title: Comparison of Orcinoside With Placebo in Treatment of MDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Kun Ming KingBio Biotechnology Co. LTD (Unknown)
Responsible Party: Principal Investigator, LI, Huafang, Executive Director of MICT, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASLST-MDD-Ⅱa-1401; 2012ZX09303-003 (Other: China National Major Project)
Record Dates: First submitted 2014-07-09; First posted 2014-07-16 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2015-03

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Orcinoside 25mg per day (Experimental)
  Interventions: Drug: Orcinoside
- Orcinoside 50mg per day (Experimental)
  Interventions: Drug: Orcinoside
- Orcinoside 100mg per day (Experimental)
  Interventions: Drug: Orcinoside
- Orcinoside 200mg per day (Experimental)
  Interventions: Drug: Orcinoside
- Orcinoside 400mg per day (Experimental)
  Interventions: Drug: Orcinoside
- Orcinoside 600mg per day (Experimental)
  Interventions: Drug: Orcinoside
- placebo (Placebo Comparator)
  Interventions: Drug: Orcinoside

INTERVENTIONS:
Drug: Orcinoside — oral, twice per day

SUMMARY:
The purpose of this study is to determine whether Orcinoside Capsule in different doses are effective in the treatment of Depression.

And to explore the preliminary information of safety and efficacy of Orcinoside Capsule in the Chinese Patients with Depression.

ELIGIBILITY:
Inclusion Criteria:

* Adult with primary diagnosis of major depressive disorder based on the criteria of DSM-IV-TR, single episode or recurrent episode, not accompanied with psychotic symptoms. Coding of diagnosis included:

296.21 MDD single episode, mild 296.22 MDD single episode, moderate 296.31 MDD recurrent episode, mild 296.32 MDD recurrent episode, moderate

* The subject is an outpatient.
* The subject is a man or woman,aged≥18 and ≤65 years.
* The total score of HAMD-17 is ≥18 and ≤24 in both screening visit and baseline visit.
* The subject is willing to take birth control measures during study period and one month after study.
* The subject understands and consents to takes part in this clinical trials. The subjects should sign informed consent.

Exclusion Criteria:

* The subject has a significant risk of suicide according to the investigator's opinion or has a score ≥3 on item 3(suicide assessment) of the HAMD or has made a suicide attempt.
* The subject has a current DSM-Ⅳ-TR axisⅠpsychiatric diagnosis other than depression.
* When the HAMD17 score of baseline visit compares with the screening visit, the decreasing rate is ≥25%.
* The subject has a current diagnosis or history of depression due to any other psychotic disorder or a general medical condition, bipolar disorder, or depression accompanied with psychotic symptoms.
* Any unstable cardiovascular, hepatic, renal, endocrine(thyroid gland dysfunction), blood,or other medical disease. Had a history of seizure disorder or other brain organic disorders.
* The subject has a diagnosis of alcohol or other substance abuse or dependence at least 1 years prior to the baseline visit.
* Known hypersensitivity to Common Curculigo Rhizome or other drugs.
* Women who were pregnant, breast-feeding, or planning to become pregnant during study. Men who have request to fertility within half of year.
* Clinically significant electrocardiographic(ECG) abnormalities or abnormal laboratory values(eg. Hepatic function above 1.5 times of clinical toplimit, renal function above toplimit, blood glucose above toplimit, cardiac troponin abnormal, thyroid gland examine index significantly abnormal).
* The subject uses antidepressant drug normally before 2 weeks of screening, and stops using psychotropic drug less than 7 half-life period (monoamine oxidase inhibitor more than 2 weeks, fluoxetine more than 1 month).
* The subject has accepted electroconvulsive therapy within 3months.
* The subject has accepted system psychotherapy within 3 months.
* The compliance of the subject is poor.
* The subject has participated in a drug clinical trial within 30 days before screening.
* The investigator think the subject is unsuitable to enrol in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03-09 (Actual); Study Completion 2016-03-09 (Actual)

PRIMARY OUTCOMES:
The change of total score from baseline in MADRS and HAMD scale | 6 weeks

SECONDARY OUTCOMES:
response rate and remission rate | 6 weeks
decreasing rate from baseline in MADRS | 6 weeks
decreasing rate from baseline in HAMD scale | 6 weeks
change from baseline in HAMA | 6 weeks
CGI(CGI-S,CGI-I) | 6 weeks
sleep VAS scale. | 6 weeks

OTHER OUTCOMES:
vital sign | 6 weeks
AE(adverse events) | 6 weeks
laboratory examination | 6 weeks
ECG | 6 weeks
C-SSRS | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Huafang LI, MD PhD, Principal Investigator — Shanghai Mental Health Center
Locations (10):
- China (10):
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Guangzhou Brain Hospital, Guangzhou, Guangdong
  - Hebei Province Mental Health Center, Baoding, Hebei
  - Wuhan Mental Health Center, Wuhan, Hubei
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - the first affiliated hospital of Xi'an Jiaotong University, Xi'an, Shan'xi
  - Xi'an Mental Health Center, Xi'an, Shan'xi
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

REFERENCES:
- [Background] Wang ZH, Huang J, Ma XC, Li GY, Ma YP, Li N, Wang JH. Phenolic glycosides from Curculigo orchioides Gaertn. Fitoterapia. 2013 Apr;86:64-9. doi: 10.1016/j.fitote.2013.01.008. Epub 2013 Jan 23. PMID 23353659